CLINICAL TRIAL: NCT05153538
Title: Evaluation of Implant Therapies Performed Under General Anesthesia in Patients With Specific Dental Needs
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2021 FAULKS Th-imp
Record Dates: First submitted 2021-11-24; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Dental Phobia; Disabilities Multiple; Complex Medical Health Condition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Implant placement is the solution of choice for replacing missing teeth in a fixed way. However, dental practitioners and surgeons are reluctant to place implants in the population of patients with special needs. They argue different arguments which involve various risk factors. A systematic review shows that it is clear that there is a gap in knowledge about implant placement in patients with special needs in order to argue the choices of prosthetic rehabilitation or abstention based on a scientific evidence-based approach. There is a need of studies with a large number of patients and implants.

The Unit of Special Care Dentistry at the University Hospital of Clermont-Ferrand started to place implants in 2007. This study should present the evaluation of the survival, success and failure rate of implants placed under general anesthesia and of the prosthesis rehabilitation that followed.

DETAILED DESCRIPTION:
Patients with special needs face multi-level barriers to dental care. Their oral health is worse than those of the general population. Delayed care in one of many reasons that lead to advanced dental disease and a need of more dental treatments. So, patients with special needs are at higher risk of early edentulism, especially since they also are at higher risk of extraction perfomed rather than conservative care. As a result, in addition to social and psychological impacts, this influences largely the oral functioning. Functional problems (mastication, swallowing) appear or are aggravated. A high prevalence of tooth loss exacerbates chewing and swallowing problems. This increases the risk of aspiration and choking, which is a major risk to general health, with bronchopulmonary disease being the leading cause of death in special needs patients. The maintenance of oral functions is therefore essential. However the conventional therapies are not adapted to patients with special needs. In particular, removable prostheses are very poorly tolerated by these patients because of the discomfort and the limitation of autonomy. The maintenance is complicated (higher prevalence of loss and repair). Many authors put forward the difficulty or even the impossibility of making removable prostheses for patients with disorders, Down's syndrome patients, patients with mental retardation or physical limitations and epileptic patients who present a risk of aspiration or ingestion of the prosthesis during seizures. In addition, the presence of associated xerostomia contraindicates the removable prosthesis and indicates the fixed solution. Implant placement is the solution of choice for replacing missing teeth in a fixed way. However, dental practitioners and surgeons are reluctant to place implants in the population of patients with special needs. They argue different arguments which involve various risk factors. A systematic review was performed to summarize the literature available about implant survival rates in patients with special needs. Twelve articles could have been included in a meta-analysis. A mean survival rate of 92% at 47,2 months on average, for an average of 23 patients and 81 implants per study was obtained. It is clear that there is a gap in knowledge about implant placement in patients with special needs in order to argue the choices of prosthetic rehabilitation or abstention based on a scientific evidence-based approach. There is a need of more studies with a large number of patients and implants.

The Unit of Special Care Dentistry at the University Hospital of Clermont-Ferrand started to place implants in 2007. This study presents the evaluation of the survival, success and failure rate of implants placed under general anesthesia and of the prosthesis rehabilitation that followed.

ELIGIBILITY:
Inclusion Criteria:

* patients from the Unit of Special Care Dentistry at the University Hospital of Clermont-Ferrand and followed in the department until the 1st of September 2021
* implants placed under general anesthesia until the 1st of September 2021

Exclusion Criteria:

* patients suffering from dental phobia with no other disability or medical health complex condition
* implants placed without the need of general anesthesia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the Unit of Special Care Dentistry at the University Hospital of Clermont-Ferrand and followed in the department until the 1st of September 2021 with implants placed by the team under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2021-12-24 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 2007 - 2021
  Informations will be seek to establish the survival rate of each implant treatment according to the Heath Scale for Dental Implants (HSDI) classification of Misch et al.
Failure rate | 2007 - 2021
  Informations will be seek to establish whether or not implants are still in the mouth

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Hospital clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No